CLINICAL TRIAL: NCT00830908
Title: An Open-Label Study of the HairMax LaserComb(r) in the Treatment of Seborrheic Dermatitis of the Scalp.
Brief Title: HairMax LaserComb Open Label Study to Treat Seborrheic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEX0903
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Seborrheic Dermatitis
Keywords: seborrheic dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LaserComb (Experimental): Patients aged 18 years and older with a diagnosis of seborrheic dermatitis of the scalp
  Interventions: Device: HairMax LaserComb

INTERVENTIONS:
Device: HairMax LaserComb — LaserComb to be used 3 times weekly on non-consecutive days, according to User Manual instructions. Use is preferably following a shower, prior to using any styling products on the hair or scalp. Hair may be wet or dry during treatment.

SUMMARY:
The purpose of this study is to test whether the stimulation of vascularization and cellular metabolism on the scalp by use of the HairMax LaserComb will produce improvement in the condition of scalp seborrheic dermatitis.

DETAILED DESCRIPTION:
This is an open label pilot study to evaluate the effects of the low-level laser light on seborrheic dermatitis of the scalp. Dandruff assessment scores for scalps with seborrheic dermatitis will be assessed at baseline with monthly evaluations during treatment, until final assessment at end of treatment at week 12.

The trial will involve 10 patients aged 18 years and older with a diagnosis of seborrheic dermatitis. Patients will use the LaserComb device three times per week on non-consecutive days for 12 weeks. No other seborrheic dermatitis products will be used during treatment. The investigator will conduct measurements of dandruff at each study visit, as a measure of efficacy.

The trial consists of 4-5 study visits (screening/baseline, week 4, week 8 and week 12). Dandruff evaluation and adverse event assessments will be performed at each visit.

Safety analysis will be assessed based on the reports of adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of seborrheic dermatitis of the scalp
* PGA of 2 (mild) or greater at baseline
* TDSS score at baseline of 2 or greater, for both scaling and inflammation
* Must agree to use of non-medicated shampoos during study period; must refrain from use of other medicated scalp products during the trial

Exclusion Criteria:

* Use of any topical or oral products that would affect assessment of the scalp SD condition, in the opinion of the primary investigator, within the following periods prior to baseline:

  * Medicated shampoos within 2 weeks of baseline
  * Topical scalp medications within 2 weeks of baseline
  * Oral medications affecting the scalp within 4 weeks of baseline
  * Other medications determined by the investigator to potentially affect the assessment of SD = washout to be determined by the investigator, as appropriate to the known medication properties
* Any current or past medical condition, including active dermatitis or any other dermatological condition, which might interfere with assessment of dandruff
* Patients using any medications that may increase photosensitivity, and thus pose a risk when undergoing LaserComb therapy
* Patients with known adverse reactions, allergy or hypersensitivity to laser light components/light sensitivity conditions
* Patients who have received any investigational drug within 30 days prior to study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a Global Outcome Score (GOS) of 0, 1 or 2 at week 12 | 12 weeks

SECONDARY OUTCOMES:
Reduction of the Total Dandruff Sum Score (TDSS) from baseline to week 12 | 12 weeks
% of subjects achieving a week 12 PGA grade of '1: slight' or '0: none' | 12 weeks
% of subjects achieving at least a 2-grade reduction in PGA from baseline to week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Gupta, M.D., Ph.D., Study Director — Mediprobe Research Inc.
Locations (1):
- Mediprobe Research Inc, London, Ontario, Canada